CLINICAL TRIAL: NCT01357122
Title: A Randomized, Observer-masked, Clinical Trial Comparing the Neusidl Corneal Inserter Corneal Transplant Technique to the Standard Forceps Insertion Technique for Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK)
Brief Title: Evaluating Results of Neusidl Corneal Inserter in Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Legacy Health System (Other)
Collaborators: Devers Eye Institute (Other); Lions Eye Bank of Oregon Vision Research Laboratory (Unknown); Fischer Surgical, Inc. (Industry)
Responsible Party: Mark A. Terry, MD/Director of Corneal Services, Deverse Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEBO-2009-1
Record Dates: First submitted 2011-05-16; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Fuchs' Corneal Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NCI Insertion (Experimental)
  Interventions: Device: NCI Insertion
- Standard Forceps Insertion (Active Comparator)
  Interventions: Procedure: Standard Forceps Insertion

INTERVENTIONS:
Device: NCI Insertion — DSAEK surgery will be performed using the NCI to insert the donor tissue.
  Arms: NCI Insertion
Procedure: Standard Forceps Insertion — DSAEK surgery will be performed using forceps to insert the donor tissue. This is our long-established technique for DSAEK, with well-documented excellent results.
  Arms: Standard Forceps Insertion

SUMMARY:
This project compares the Neusidl Corneal Injector (NCI) device developed by Fischer Surgical, Inc. for the delivery of tissue into the eye in DSAEK surgery to the current standard forceps insertion DSAEK technique. The goal of this study is to examine the damage to the corneal endothelium resulting from the use of the NCI device in comparison to the use of our standard surgical DSAEK technique over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and over
* A diagnosis of Fuchs' Corneal Endothelial Dystrophy

Exclusion Criteria:

* Under age 21
* Diagnosis of advanced glaucomatous disease
* Diagnosis of significant retinal disease
* Diagnosis of any other corneal dystrophy
* Previous corneal transplant surgery
* Previous glaucoma surgery
* Previous retinal surgery
* Previous refractive surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Decrease in Endothelial Cell Density From Baseline Over Time | 6, 12, 24, and 60 Months
  Endothelial cell density (ECD) will be captured at each follow-up visit using a non-contact specular microscope. % Cell reduction from pre-operative baseline ECD will be calculated for each patient, and compared between treatment arms to evaluate each instrument's effect on long-term post-operative endothelial cell density.

SECONDARY OUTCOMES:
Adverse events | Any time during follow-up period (5 years)
  Each patient will be monitored for incidence of graft dislocation, primary graft failure, immunologic graft rejection, and late endothelial failure. Rates will be compared between groups to ensure that the NCI does not increase the risk of these adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Terry, MD, Principal Investigator — Devers Eye Institute
Locations (1):
- Devers Eye Institute, Portland, Oregon, United States